CLINICAL TRIAL: NCT00891384
Title: A Randomised Comparison of Daily 25 mg Versus 5 mg Lenalidomide as Maintenance Therapy After High-dose Therapy and Autologous Stem Cell Transplantation in Patients With Multiple Myeloma
Brief Title: Comparison of 25mg Versus 5 mg Lenalidomide as Maintenance Therapy in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LenaMain-Trial
Record Dates: First submitted 2009-04-24; First posted 2009-05-01 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; maintenance therapy; lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 25 mg lenalidomide
  Interventions: Drug: Lenalidomide
- 2 (Experimental): 5 mg lenalidomide
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Patients will receive maintenance therapy according to their assigned treatment arm: 25 mg daily for 21 days every 28 days. During the treatment period patients will be seen every 4 weeks until disease progression is documented. All patients who have to discontinue the study drug will be followed until disease progression.
  Other Names: Revlimid
  Arms: 1
Drug: Lenalidomide — Patients will receive maintenance therapy according to their assigned treatment arm:5 mg daily for 21 days every 28 days. During the treatment period patients will be seen every 4 weeks until disease progression is documented. All patients who have to discontinue the study drug will be followed until disease progression
  Other Names: Revlimid
  Arms: 2

SUMMARY:
This trial is a randomised, parallel-group, multicenter phase III study for maintenance therapy with lenalidomide in patients with multiple myeloma who were treated with high-dose therapy and autologous stem cell transplantation as first line therapy.

DETAILED DESCRIPTION:
High-dose therapy will be performed as first line treatment. After high-dose therapy and autologous stem cell transplantation the patients will be included and randomised. Three month after high-dose therapy all patients will receive consolidation therapy with 6 cycles of lenalidomide 25 mg daily for 21 days every 28 days. Afterwards patients will receive maintenance therapy according to their assigned treatment arm. Randomisation will be performed in a 1:1 ratio to continuous maintenance therapy with either 25mg or 5mg lenalidomide daily for 21 days every 28 days.Randomisation will be stratified by ISS-stage (1+2 vs 3, age (younger than 66 years versus 66 years or older), response after high-dose therapy (CR+vgPR vs PR vs MR/SD. Patients will be treated until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age 18-75 years
* Able to adhere to the study visit schedule and other protocol requirements
* Patients with multiple myeloma who have received high-dose therapy and autologous stem cell transplantation as first-line therapy within the last 90 - 120 days and have not shown progressive disease afterwards.
* Patients may have received up to 6 cycles of prior induction therapy and up to 2 cycles of prior mobilisation chemotherapy. A bortezomib or thalidomide induction therapy is allowed. Patients may also have received prior radiation therapy
* Measurable levels of myeloma paraprotein in serum (>0.5 g/dL) or urine (>0.2 g/24hours) or measurable free light chains (FLC) in serum (>50 mg/l) with an abnormal FLC ratio must be documented at the time of first diagnosis.
* ECOG performance status = 2 at study entry
* Laboratory and functional test results within these ranges:

  * ANC ≥ 1,000/μL
  * Platelet count ≥ 100,000/μL
  * Total bilirubin 2.5 mg/dL
  * AST (SGOT) and ALT (SGPT) 3 x ULN
  * Patients with impaired renal function can be included
* The patient must be able to adhere to the pregnancy precautions
* Disease free of prior malignancies for 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females
* Any condition or laboratory abnormality which places the subject at an unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Known allergic/hypersensitivity reaction to thalidomide, lenalidomide or any components of the treatment
* Any cutaneous grade ≥ 3 adverse reaction (for example desquamating rash) while taking thalidomide or similar drugs
* Any prior use of lenalidomide
* Known positive for HIV or active infectious hepatitis, type A, B or C

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
event-free survival | 6 years

SECONDARY OUTCOMES:
safety, tolerability and feasibility | 6 month
Improvement of remission rate | 6 years
evaluate quality of life | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Guido Kobbe, PD Dr., Principal Investigator — Departement of Hematology, Oncology and Clinical Immunology
Locations (5):
- Germany (5):
  - Medizinische Klinik, Abteilung Innere Medizin, Heidelberg, Baden-Wurttemberg
  - Clinic of Justus-Liebig-University, Medical Clinic for Hematology and Medical Oncology, Giessen, Hesse
  - St. Johannes Hospital, Medical Clinic II, Duisburg, Northwest
  - Departement of Hematology, Oncology and Clinical Immunology, Düsseldorf, Northwest
  - Bone Marrow Transplantation Unit, University Hospital Hamburg-Eppendorf, Hamburg